CLINICAL TRIAL: NCT04947670
Title: A Prospective, Multicenter, Randomized, Blinded, Sham-controlled, Feasibility Study of Renal Denervation in Patients With Chronic Heart Failure
Acronym: RE-ADAPT-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment problems
Sponsor: Universität des Saarlandes (Other)
Collaborators: Interdisciplinary Center Clinical Trials (IZKS), University Medical Center Mainz (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RE-ADAPT-HF (2021)
Record Dates: First submitted 2021-06-24; First posted 2021-07-01 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic Heart Failure; Cardio-Renal Syndrome
MeSH Terms: conditions — Cardio-Renal Syndrome

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double-blind, sham-controlled, multicenter, feasibility study. Patients will be screened for meeting eligibility and centrally randomized to receive either renal denervation or sham procedure. Best medical therapy will be provided to all patients. Optional cross-over after 12 months for sham-group patients. Thus, there is an intra-individual control in patients of the control group and all of the randomized patients are entitled to receive study treatment.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Unblinded interventionist, unblinded intervention team and blinded study team at each center, blinded patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Renal denervation and maintenance of heart failure medications
  Interventions: Procedure: Renal arteriography followed by renal denervation
- Control Group (Sham Comparator): Sham intervention, maintenance of heart failure medications with option for cross-over renal denervation treatment after 12 months
  Interventions: Procedure: Sham Renal arteriography

INTERVENTIONS:
Procedure: Renal arteriography followed by renal denervation — Renal arteriography followed by renal denervation
  Arms: Treatment Group
Procedure: Sham Renal arteriography — Renal arteriography only
  Arms: Control Group

SUMMARY:
The renin-angiotensin-aldosterone axis has been found to be a key system involved in heart failure disease progression and it may be inhibited by renal sympathetic denervation. Therefore, a clear need exists for further strategies to beneficially manipulate the sympathetic activation that is characteristic of the heart failure disease process.

The combined experience in the pilot studies and the EU randomized, controlled study indicates that the Paradise Catheter System can safely denervate renal sympathetic nerves of the kidney without significant periprocedural complications.

Preliminary results of a pilot study of catheter-based renal denervation in a small number of CHF patients did not show evidence of safety issues but suggest improvements in CHF symptoms. This trial will explore the safety and feasibility of renal denervation in a significantly higher number of patients with chronic heart failure. Both inter-individual and intra-individual controls will be used in order to obtain sufficient data and to in order to enable both treatment and control group to receive renal denervation.

Additionally, this feasibility trial to describe the safety and feasibility of renal denervation in patients with elevated sympathetic activity as in patients with chronic heart failure, will further the understanding of the role of renal nerves in the control of chronic heart failure and the pathogenesis of both ventricular remodeling and cardio-renal syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patient with CHF diagnosed for at least 3 months prior to consent
* 6-min walk distance ≤350 m
* NYHA Class II-III symptoms of CHF
* Systolic left ventricular dysfunction as assessed by echocardiogram with left ventricular ejection fraction <45%
* eGFR calculated (CKD-EPI) >30 ml/min/1.73 m2
* NT-pro-BNP >450 pg/ml, >900 pg/ml for patients with atrial fibrillation
* Optimal medical drug therapy according to current guidelines for CHF management. This medication may include loop diuretics, ACEi/ARBs, ARNI, SGLT-2 inhibitors, aldosterone antagonists, and beta-blockers, unless intolerance to any of the above is documented. Treatment for HF must be stable (including drug and dose) for 4 weeks prior to randomization, except diuretics (2 weeks stable)
* Appropriate use of medical devices such as an implantable cardioverter defibrillator (ICD) or a cardiac resynchronization therapy (CRT) consistent with prevailing local or international guidelines, and if a device is required, it must have been implanted for at least 3 months prior to consent for CRT and 1 month prior to consent for ICD
* Age ≥18 years and ≤80 years

Exclusion Criteria:

* Renal arterial anatomy that is ineligible for treatment
* Myocardial infarction, unstable angina pectoris, or a cerebrovascular accident within 12 weeks prior to consent
* Office systolic BP at screening <90 mmHg
* Clinically significant cardiac structural valvular disease, unless corrected by a properly functional prosthetic valve
* Hypertrophic obstructive cardiomyopathy
* Major surgery in the previous 12 weeks prior to consent
* Hospitalization for decompensated CHF in the <30 days prior to consent
* Parenteral therapy for the treatment of CHF
* Respiratory support (excluding sleep apnea therapy)
* Left ventricular assist or planned heart transplantation
* Patient is pregnant, nursing, or planning to be pregnant
* Ineligibility to consent
* Primary pulmonary hypertension (systolic PAP >70 mmHg)
* BMI ≥40 kg/m²
* Any condition that would contraindicate the assessment of 6-min walk distance.
* Patient has type I diabetes mellitus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
6 Minute Walk Test | 6 months
  Change in 6-min walk distance

SECONDARY OUTCOMES:
NT-proBNP | 6 months
  Change in plasma NT-proBNP values
KCCQ | 6 months
  Change in Overall Summary Score measured by Kansas City Cardiomyopathy Questionnaire (KCCQ)
EQ-5D | 6 months
  Change in Chronic Heart Failure Questionnaire Self-Administered Standardized format (CHQ-SAS) dyspnea score
eGFR | 6 months
  chronic eGFR slope defined as eCRF

CONTACTS AND LOCATIONS:
Overall Officials: Felix Mahfoud, MD, Principal Investigator — Saarland University Medical Center
Locations (1):
- Saarland University Medical Center, Department for Internal Medicine III, Homburg/Saar, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No